CLINICAL TRIAL: NCT00817531
Title: A Biologic Efficacy Study of Dasatinib, a Multi-Targeted Tyrosine Kinase, in Locally Advanced Triple-Negative Breast Cancer Patients Developing Effective Therapies for Er-Negative Breast Cancer Using Genomics and Proteomics: Project 3
Brief Title: Efficacy Study of Dasatinib in Locally Advanced Triple-Negative Breast Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated due to futility after interim analysis
Sponsor: Baylor Breast Care Center (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H 21592
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Results first posted 2012-07-17 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All subjects take open label Dasatinib (Experimental): Dasatinib / Sprycel 100 mg
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — pill form, 100 mg daily
  Other Names: Sprycel

SUMMARY:
We want to learn if dasatinib will make triple negative breast cancers smaller. We also hope that we can learn more about what makes triple negative breast cancers grow. We believe this information will help us to predict which patients will benefit from taking this drug or other drugs like it.

This study is a "neoadjuvant study", which means that it is only open to women who have not had any treatment for their breast cancer. Neoadjuvant studies allow the study doctor to look at how the cells in your cancer change after taking the study medication. This will help us to understand whether or not dasatinib is an effective treatment for breast cancer. It will also help us to learn more about triple negative breast cancer and how to treat it.

DETAILED DESCRIPTION:
Women who have been recently diagnosed with a type of breast cancer called "triple negative", and have not yet received any type of treatment (surgery, radiation therapy, etc.) for breast cancer are among the patient population this study will seek. "Triple negative" means breast cancer is not estrogen receptor positive (ER+), progesterone receptor positive (PgR+) or human epidermal growth factor receptor positive (HER2+). Some types of breast cancers "overexpress" one or more of these receptors. "Overexpress" means that the cancer cells have too many of these receptors. ER and PgR are hormone receptors that are located on some types of breast cancer cells. When these receptors are present, the hormones estrogen and progesterone are able to tell cancer cells to grow and divide.

This kind of breast cancer does not have an over-production (overexpression) of these three receptors, and that is why we call it "triple-negative" breast cancer.

We are trying to find new and better treatments for women with triple negative breast cancer. We do not know what causes triple negative breast cancers to grow. Other research studies have shown that "triple negative" breast cancers overexpress different types of receptors. These receptors might help the cancer to grow.

We will be testing a drug called dasatinib. Dasatinib is a drug that is made by Bristol-Myers Squibb. It is sold under the name of Sprycel. It was first used to treat patients with leukemia, a type of blood cancer.

Dasatinib interferes with the growth of some cancers. Dasatinib attaches to the cancer cell and slows down or stops the cancer cell from growing. It is approved by the Food and Drug Administration (FDA), but not for the kind of cancer that you have been diagnosed with.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with triple negative breast cancer (breast cancer is not estrogen receptor positive (ER+), progesterone receptor positive (PgR+) or human epidermal growth factor receptor positive (HER2+)

  1. Clinical stage II or stage III invasive mammary carcinoma, confirmed by histological analysis, as defined in the study protocol.
  2. Subject's age must be greater than or equal to 18 years.
  3. ECOG Performance Status of 0-1.
  4. Subjects must have measurable* tumor at the primary site. *Measurable disease is defined as follows: Any mass that can be reproducibly measured by physical examination, mammogram, and/or ultrasound and can be accurately measured in at least one dimension (longest diameter to be recorded) as 10 mm (1 cm).
  5. No history of prior chemotherapy for primary breast cancer.
  6. Patients with a prior history of contralateral breast cancer are eligible if they have no evidence of recurrence of their initial primary breast cancer within the past 5 years.
  7. Women may have been taking tamoxifen or raloxifene as a preventive agent prior to study entry but must have discontinued the drug for at least 21 days prior to study enrollment.
  8. Adequate organ function, as defined by the following: a) Total bilirubin < 2.0 times the institutional Upper Limit of Normal (ULN) b) Hepatic enzymes (AST, ALT ) ≤ 2.5 times the institutional ULN c) Serum sodium, potassium, magnesium, phosphate, and calcium levels greater than or equal to the Lower Limit of Normal (LLN). d) Serum Creatinine < 1.5 time the institutional ULN e) Hemoglobin, Neutrophil count, Platelets, PT, PTT all Grade 0-1, as defined by the NCI CTCAE v3.0.
  9. Ability to swallow and retain oral medications (dasatinib must be swallowed whole).
  10. Subject must not be taking any prohibited medications, as defined in Section 6.5 of the study protocol.
  11. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (sensitivity < 25 IU/L) within 72 hours prior to beginning study medication.
  12. WOCBP must agree to utilize an adequate method of contraception throughout treatment, and for at least 4 weeks after stopping study medication. 13. Signed, written informed consent, including a HIPAA form, as per institutional guidelines.

Exclusion Criteria:

1. Locally recurrent breast cancer.
2. History of prior chemotherapy for breast cancer.
3. History of malignancy requiring radiotherapy or systemic treatment within the past 5 years.
4. Presence of any concurrent medical condition that would increase the risk of toxicity, including the following: •Pleural or pericardial effusion of any grade •Uncontrolled angina •Congestive heart failure •Myocardial infarction within the past 6 months •Diagnosed congenital long QT syndrome •Any history of clinical significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes) •Prolonged QTc interval (> 450 ms) on pre-study ECG •Uncorrectable hypokalemia or hypomagnesia •Significant bleeding disorder unrelated to cancer, including: - History of congenital bleeding disorders (e.g. von Willebrand's disease) - Acquired bleeding disorder that has been diagnosed within the past year (e.g. acquired anti-factor VIII antibodies) - Ongoing or recent (less than or equal to 3 months) significant gastrointestinal bleeding.
5. Subjects taking any prohibited medications will be excluded from study, as defined in Section 6.5 of the study protocol.
6. WOCBP who are pregnant or breastfeeding or who are unwilling to use an acceptable method of contraception for the duration of study therapy and for at least 4 weeks after cessation of study drug.
7. Active or uncontrolled infection.
8. Dementia, altered mental status, or any psychiatric condition that would prohibit the understanding or rendering of informed consent.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar Rimawi, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Lester and Sue Smith Breast Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started recruitment in December 2010. Baylor college of Medicine is the only site of the study.
Pre-assignment Details: each patient have to be eligible and pass all screening tests after signing the consent to be enrolled in the study.
Groups:
- Dasatinib: Patients took Dasatinib 100mg daily
Period: Overall Study
Arm/Group | Dasatinib
Started | 22 (22 patients were eligible for this study and started the treatment.)
Completed | 20 (20 out of 22 patients finished study treatment. 2 patients stopped the treatment after the 1st week.)
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 48.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Clinical Efficacy
Description: The clinical response was assessed using RECIST and based on the changes in the longest diameter of the target lesion measured. Complete Response (CR), Disappearance of the target lesion; Partial Response (PR), >=30% decrease in the diameter of target lesion compared to baseline; Progressive disease (PD), >= 20% increase in the diameter of target lession, taking as reference the smallest diameter recorded since the baseline measurement or the appearance of new lesion; Stable disease (SD), neither sufficient shrinkage as PR or sufficient increase as PD.
Time Frame: Assessment at pre-surgery or 3 to 4 weeks of treatment.
Population: All patients started the treatment will be included in the analysis
Measure: Number; unit: participants
Groups:
- Dasatinib: Dasatinib 100 mg once daily
Arm/Group | Dasatinib
Number analyzed (Participants) | 22
participants
  Partial Response (PR) | 2
  Stable Disease (SD) | 15
  Progression Disease (PD) | 5

ADVERSE EVENTS:
Time Frame: 3-4 weeks
Description: Following the patient's written consent to participate in the study, then to the end of 3-4 week treatment
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=22)
Cardiac infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=22)
ALT, SGPT(serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 9 (10)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 11 (12)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4 (4)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 5 (5)
Hemoglobin (Blood and lymphatic system disorders) | 6 (6)
Infection (Infections and infestations) | 3 (4)
Nausea (Gastrointestinal disorders) | 4 (5)
Pain (General disorders) | 15 (17)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 (4)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 2 (3)

LIMITATIONS AND CAVEATS:
The study was terminated after internal analysis due to treatment futility. It does not meet the required number of responses to continue the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes